CLINICAL TRIAL: NCT03271385
Title: EARLY Differentiation of MYOcardial Hypertrophy Between Hypertensive Heart Disease and Hypertrophic Cardiomyopathy
Brief Title: Differentiation HHD From HCM (EARLY-MYO-HHD)
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Ruijin Hospital (Other); LanZhou University (Other); Kunming Medical University (Other); Beijing Anzhen Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20170406J
Record Dates: First submitted 2017-08-21; First posted 2017-09-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2021-09

CONDITIONS: Hypertrophic Cardiomyopathy; Hypertensive Heart Disease
Keywords: hypertrophic Cardiomyopathy; hypertensive Heart Disease; cardiac magnetic resonance
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hypertrophic cardiomyopathy group: The hypertrophic cardiomyopathy was diagnosed by left ventricular hypertrophy via echocardiography (wall thickness >15 mm) with either genetic determination of a pathogenic mutation or ) left ventricular hypertrophy (LVH) (end-diastolic wall thickness >15 mm) with resting left ventricular outflow tract obstruction or hypertrophy in a recognisable pattern, i.e., ventricular bulge in apical-variant HCM. And then patients with hypertrophic cardiomyopathy were evaluated by the predetermined differentiating formula.
  Interventions: Diagnostic Test: evaluated by the predetermined differentiating formula
- hypertensive heart disease group: The diagnosis of hypertensive heart disease was based on medical history and conventional echocardiography. Long durations of uncontrolled hypertension for at least 5 years with systolic blood pressure [BP] ≥150 mm Hg or diastolic BP ≥90 mm Hg or both in the absence of other cardiac or systemic diseases were used as criteria. And then patients with hypertensive heart disease were evaluated by the predetermined differentiating formula.
  Interventions: Diagnostic Test: evaluated by the predetermined differentiating formula
- control group: The healthy age-matched controls were generally volunteers with a normal electrocardiogram, normal echocardiographic examination, and overall normal CMR findings. And then patients with normal findings were were evaluated by the predetermined differentiating formula.
  Interventions: Diagnostic Test: evaluated by the predetermined differentiating formula

INTERVENTIONS:
Diagnostic Test: evaluated by the predetermined differentiating formula — After recruiting patients, collecting the baseline data, a CMR scan will be carried out and post-processed, a predetermined differentiating formula (including left ventricular morphology, ejection fraction, presence of late gadolinium enhancement, T1 value and strain data) will be used to produce a cardiac values, which is to be input into our differentiating flow.

SUMMARY:
Differentiating hypertrophic cardiomyopathy (HCM) from hypertensive heart disease (HHD) unavoidably encounters diagnostic challenges especially in patient of suspected HCM with history of hypertension. Diverse and overlapping forms of HCM can often lead to ambiguity when diagnosis is based on a single genetic or morphological index.

The investigators have deduced a integrated formula based on cardiac magnetic resonance (CMR) imaging and established a differentiating flow-chart between HCM and HHD, the investigators aim to identify their method in the current multi-center trial.

DETAILED DESCRIPTION:
Both hypertrophic cardiomyopathy (HCM) and hypertensive heart disease (HHD) present left ventricular hypertrophy (LVH), but the prognosis varies. Nevertheless, the feasibility of distinguishing these two conditions is limited by the fact that overlapping LVH and diverse forms of HCM can often lead to diagnostic ambiguity when diagnosis is based on a single morphological index. Diagnosis is more difficult in a patient with a history of hypertension and with left ventricular wall thickness between 11 and 15 mm. It also puzzles the situation when hypertrophy without outflow-track obstruction was found in hypertensive subjects which might not be explained solely by the history of hypertension.

The investigators have deduced an integrated formula based on cardiac magnetic resonance (CMR) imaging and established a differentiating flow-chart between HCM and HHD. In this study, the investigators aim to explore the applicability of the quantifying scheme for distinguishing HCM from HHD in the multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

1. Control group: (1) Absence of known systemic diseases; (2)Normal examinations（normal findings in both echocardiography and CMR）.
2. Hypertrophic cardiomyopathy: 1) genetic determination of a pathogenic mutation or 2) left ventricular hypertrophy (LVH) (end-diastolic wall thickness >15 mm) with resting left ventricular outflow tract obstruction or 3) hypertrophy in a recognizable pattern, i.e., ventricular bulge in apical-variant HCM; Of note, patients with documented HCM were divided into subgroups based on whether concomitant with hypertension or left ventricular outflow tract (LVOT) obstruction.
3. Hypertensive Heart Disease: (1) Long durations of uncontrolled hypertension (systolic blood pressure≥150 mm Hg or diastolic blood pressure ≥90 mm Hg); Echocardiography: left ventricular wall thickness in diastolic >11mm; Absence of other cardiac or systemic diseases; (2) left ventricular mass/body surface area >115 g/m2 (Male) or >95 g/m2 (Female).

Exclusion Criteria:

1. Documented coronary artery disease: previous history or CAG>50%;
2. NYHA Ⅳ level;
3. Severe aortic valve stenosis;
4. Standard metallic contraindications to CMR;
5. Systemic diseases or Infiltrative cardiomyopathy;
6. Septal ablation for drug-refractory hypertrophic obstructive cardiomyopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects were prospectively enrolled into 3 cohorts between July 2017 and June 2020. The cohorts were divided as follows: the hypertrophic cardiomyopathy, hypertensive heart disease and control groups
Sampling Method: Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
validation of the algorithm in all patients | after post-procession and complete the flow chart within 24 hours
  Evaluate the area under the curve of our algorithm compared with single parameter (wall thickness, strain) in all patients

SECONDARY OUTCOMES:
validation of the algorithm in subgroup patients | after post-procession and complete the flow chart within 24 hours
  Evaluate the area under the curve of our algorithm compared with single parameter (wall thickness, strain) in subgroup patients (HHD and HCM/HBP-; HHD and HCM/HBP+; HHD and HCM/OBSR-; HHD and HCM/HBP+/OBSR-)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiaotong University; Lianming Wu, MD, Study Director — RenJi Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No